CLINICAL TRIAL: NCT00083486
Title: Treatment of Anemia in Patients With Cancer Who Are Not Currently Receiving Chemotherapy or Radiotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Purpose: Treatment
Other Study IDs: CR010939; EPO-CAN-203
Record Dates: First submitted 2004-05-24; First posted 2004-05-27 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2011-04

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to determine the effectiveness of different doses of epoetin alfa for treating anemia in patients who have cancer; or patients who no longer have any signs of cancer, but remain anemic as a result of their treatment. These patients should not be currently receiving chemotherapy or radiotherapy. A subject's participation in the study will last approximately 6 months. Subjects will receive weekly doses of epoetin alfa or placebo. Their hemoglobin will be tested every week.

ELIGIBILITY:
Inclusion Criteria:

* Body weight >/=99 lbs
* ECOG 0-2
* Anemia results from cancer, chemotherapy, radiotherapy or an association with hormonal therapy or immunotherapy
* Screening hemoglobin level of </=11.0 g/dL for men or </=10.0 for women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-02; Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Heritage Physician Group-Oncology, Hot Springs, Arkansas
  - Spalding Oncology Services, Griffin, Georgia
  - Southern Illinois Hematology, Centralia, Illinois
  - BioLab Research, Rockville, Maryland
  - Slocum-Dickson Medical Group, PC, New Hartford, New York
  - NorthEast Urology Research, Concord, North Carolina
  - Mid Ohio Oncology Hematology, Columbus, Ohio
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Caroline Cancer Center, Aiken, South Carolina
  - Charleston Hematology Oncology, Charleston, South Carolina
  - Charleston Cancer Care, Charleston, South Carolina
  - Volunteer Research Group, Knoxville, Tennessee